CLINICAL TRIAL: NCT06699979
Title: Comprehensive Multi-Omics Analysis of Early-Stage Lung Cancer Exhibiting Distinct Phenotypes
Brief Title: Multi-omics Study of Early-stage Lung Cancer with Distinct Phenotypes
Status: Recruiting | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Chen Chen, Associate Professor, Second Xiangya Hospital of Central South University
Other Study IDs: LYEC2024-0320
Record Dates: First submitted 2024-11-09; First posted 2024-11-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer Associated with Cystic Airspaces; Multiple Primary Lung Cancers; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh tumor tissue, adjacent normal tissue, peripheral blood cells, and plasma samples were collected from each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Non-small cell lung cancer: Early-stage lung cancer exhibiting distinct phenotypes including lung cancer associated with cystic airspaces, multiple primary lung cancers, and so on.

SUMMARY:
The goal of this observational study is to investigate the multi-omics characterization early-stage lung cancer exhibiting distinct phenotypes including lung cancer associated with cystic airspaces, multiple primary lung cancers, and so on. The main questions it aims to answer are:

* What are the differences in pathogenesis of non-small cell lung cancer with different phenotypes explored by multi-omics?
* Whether differential genes lead to potential prognostic models and therapeutic targets? Participants will be followed up after surgery to answer prognosis: whether they have recurred, and the time to recurrence.

ELIGIBILITY:
Cohort 1: Multi-omics study in early-stage synchronous multiple primary lung cancer

Inclusion criteria:

1. Male or female patients:18-75 years old;
2. ECOG score:0-1;
3. Histopathologically confirmed TNM stage I-II NSCLC;
4. Considered multiple or solitary primary lung cancer by clinical criteria (Martini-Melamed criteria and ACCP criteria);
5. Good compliance, family members agree to cooperate to receive survival follow-up;
6. Understand and voluntarily sign the informed consent.

Exclusion criteria:

1. A history of previous or co-existing malignant tumors;
2. Systemic anti-tumor therapies, including chemotherapy, radiotherapy, or targeted therapies (such as monoclonal antibodies, small-molecule tyrosine kinase inhibitors, among others), were administered prior to enrollment;
3. Refusal to participate in the study.

Cohort 2: Multi-omics study of lung cancer associated with cystic airspaces

Inclusion criteria:

1. Male or female patients:18-75 years old;
2. ECOG score:0-1;
3. Histopathologically confirmed TNM stage I-II NSCLC;
4. CT findings show solitary or multiple nodules with cystic airspaces.

Exclusion criteria:

1. A history of previous or co-existing malignant tumors;
2. Systemic anti-tumor therapies, including chemotherapy, radiotherapy, or targeted therapies (such as monoclonal antibodies, small-molecule tyrosine kinase inhibitors, among others), were administered prior to enrollment;
3. Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer with indication for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Immune repertoire sequencing | From enrollment to the end of surgery for 3 years
DNA methylome sequencing | From enrollment to the end of surgery for 3 years
RNA sequencing | From enrollment to the end of surgery for 3 years

SECONDARY OUTCOMES:
Genomic sequencing | From enrollment to the end of surgery for 3 years
Metabolomics analysis | From enrollment to the end of surgery for 3 years
Radiomics analysis | From enrollment to the end of surgery for 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhong WZ, Wang Q, Mao WM, Xu ST, Wu L, Shen Y, Liu YY, Chen C, Cheng Y, Xu L, Wang J, Fei K, Li XF, Li J, Huang C, Liu ZD, Xu S, Chen KN, Xu SD, Liu LX, Yu P, Wang BH, Ma HT, Yan HH, Yang XN, Zhou Q, Wu YL; ADJUVANT investigators. Gefitinib versus vinorelbine plus cisplatin as adjuvant treatment for stage II-IIIA (N1-N2) EGFR-mutant NSCLC (ADJUVANT/CTONG1104): a randomised, open-label, phase 3 study. Lancet Oncol. 2018 Jan;19(1):139-148. doi: 10.1016/S1470-2045(17)30729-5. Epub 2017 Nov 21. PMID 29174310